CLINICAL TRIAL: NCT07370844
Title: A Prospective Randomized Controlled Trial of VR Training to Improve Postoperative Cognitive Function in Elderly Patients With Cerebral Small Vessel Disease Undergoing Non-Cardiac Surgery
Brief Title: VR Training to Improve Postoperative Cognitive Function in Elderly Patients With Cerebral Small Vessel Disease Undergoing Non-Cardiac Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Peking University First Hospital (Other); Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Li Zhengqian, Associate Chief Physician, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TY2025014
Record Dates: First submitted 2026-01-14; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Small Vessel Disease; Postoperative Cognitive Function
Keywords: Cerebral Small Vessel Disease; Postoperative Cognitive Function; Postoperative Delirium; Virtual Reality
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Emergence Delirium

STUDY DESIGN:
Intervention Model Description: A third-party statistician generated the allocation sequence using R 4.3.3 with a dynamic block design (mixed block sizes of 4 and 6), stratified by study site; the randomization scheme was uploaded to the REDCap system, where patient eligibility was verified before enrollment, and upon entering patient data into REDCap, the system automatically executed the stratified randomization.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative Training Group (Experimental)
  Interventions: Device: Virtual reality cognitive function training
- Preoperative Non-Training Group (Sham Comparator)
  Interventions: Device: Virtual scene intervention

INTERVENTIONS:
Device: Virtual reality cognitive function training — Participants will receive VR-based cognitive training over 4-5 days prior to surgery, with three daily 30-minute sessions (8:00-10:00 AM, 12:00-2:00 PM, and 5:00-7:00 PM), ensuring a total preoperative training duration ≥6 hours. The intervention utilizes an immersive VR environment that simulates real-world scenarios and tasks. Training modules target multiple cognitive domains, including memory, executive function, calculation, and abstract reasoning, designed as engaging, game-like activities with a gradual learning curve. Each participant's regimen is personalized based on baseline cognitive assessments or physician prescriptions, adhering to the "6-hour rule" for standardized efficacy evaluation. The system incorporates adaptive difficulty adjustment, dynamically modifying task complexity in response to real-time performance.
  Arms: Preoperative Training Group
Device: Virtual scene intervention — The control group will receive non-interactive VR exposure using identical equipment and session duration as the training group (3×30-minute daily sessions for 4-5 days, totaling ≥6 hours), with all interactive functions disabled to eliminate potential media-related biases (e.g., 2D/3D cognitive load differences from tablet-based interventions) and ensure between-group differences stem solely from interactive training while maintaining blinding integrity through equivalent hardware deployment.
  Arms: Preoperative Non-Training Group

SUMMARY:
This clinical study aims to investigate whether virtual reality (VR)-based cognitive training can help improve postoperative cognitive function in elderly non-cardiac surgery patients with pre-existing cerebral small vessel disease (CSVD). As the global aging population undergoes an increasing number of surgical procedures, perioperative neurocognitive disorders (PND) have emerged as a serious complication among surgical patients, potentially prolonging hospital stays and increasing the risk of developing Alzheimer's disease. The study employs an innovative VR system that integrates eye-tracking cognitive assessment with interactive rehabilitation games to evaluate and train patients' cognitive function prior to non-cardiac and non-cranial surgeries. Conducted at Peking University Third Hospital, Peking University First Hospital, and Xuanwu Hospital of Capital Medical University, this research specifically targets patients undergoing general surgery, orthopedic surgery, and other non-cranial/non-cardiac procedures. It seeks to validate whether this technology-based intervention can effectively enhance postoperative cognitive function in this population while exploring its underlying mechanisms. The findings may offer a practical solution for protecting cognitive health in elderly patients during recovery from routine surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥60;
2. Preoperative MRI-confirmed cerebral small vessel disease;
3. Scheduled to undergo non-cardiac, non-craniotomy procedures under general anesthesia;
4. ASA physical status classification: I-III;
5. No use of cognitive-enhancing medications within 3 months prior to surgery;
6. Voluntary participation with signed informed consent

Exclusion Criteria:

1. Contraindications to cranial MRI (e.g., cardiac pacemaker, metallic implants, etc.);
2. Intolerance to VR equipment during pre-training adaptation (e.g., dizziness, nausea, vomiting, or other subjective discomfort);
3. Severe visual or auditory impairment;
4. Severe hepatic or renal dysfunction;
5. Pre-existing neuropsychiatric disorders (e.g., schizophrenia, epilepsy, Parkinson's disease, or active delirium);
6. Inability to complete preoperative neuropsychological assessments (e.g., dementia, deaf-mutism, or communication barriers);
7. Use of sedatives, antidepressants, or history of psychoactive substance abuse/alcoholism

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in postoperative cognitive score from baseline | At admission, on postoperative day 5 (or before discharge), and at 1, 6, and 12 months postoperatively
  Trained research personnel (certified by neurologists) administer the Montreal Cognitive Assessment (MoCA) to evaluate eight cognitive domains (visuospatial ability, executive function, memory, attention, calculation, language, abstract thinking, and orientation), with total scores ranging 0-30 (normal cognition defined as ≥26).We defined an increase in MoCA of ≥ 2 points as cognitive improvement

SECONDARY OUTCOMES:
Occurrence of postoperative delirium | From the first day to the fifth day after surgery or from the first day after surgery to before discharge
  Follow up personnel use the Confusion Assessment Method(CAM) scale to evaluate the occurrence of postoperative delirium after anesthesia surgery
Amplitude of Low-Frequency Fluctuation（ALFF） of brain regions | At enrollment and immediately after completion of the preoperative intervention
  Blood Oxygen Level Dependent Functional Magnetic Resonance Imaging (BOLD-fMRI) was used to measure changes in brain regions activation
Fractional Amplitude of Low-Frequency Fluctuation（fALFF) of brain regions | At enrollment and immediately after completion of the preoperative intervention
  Blood Oxygen Level Dependent Functional Magnetic Resonance Imaging (BOLD-fMRI) was used to measure changes in brain regions activation
Regional Homogeneity（ReHo） of brain regions | At enrollment and immediately after completion of the preoperative intervention
  Blood Oxygen Level Dependent Functional Magnetic Resonance Imaging (BOLD-fMRI) was used to assess the synchronization of neuronal activity within brain regions

CONTACTS AND LOCATIONS:
Overall Officials: Zhengqian Li, Principal Investigator, Principal Investigator — Peking University Third Hospital
Locations (3):
- China (3):
  - Peking University First Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Xuanwu Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Chen CC, Li HC, Liang JT, Lai IR, Purnomo JDT, Yang YT, Lin BR, Huang J, Yang CY, Tien YW, Chen CN, Lin MT, Huang GH, Inouye SK. Effect of a Modified Hospital Elder Life Program on Delirium and Length of Hospital Stay in Patients Undergoing Abdominal Surgery: A Cluster Randomized Clinical Trial. JAMA Surg. 2017 Sep 1;152(9):827-834. doi: 10.1001/jamasurg.2017.1083. PMID 28538964
- [Result] de Vries NM, Staal JB, van der Wees PJ, Adang EM, Akkermans R, Olde Rikkert MG, Nijhuis-van der Sanden MW. Patient-centred physical therapy is (cost-) effective in increasing physical activity and reducing frailty in older adults with mobility problems: a randomized controlled trial with 6 months follow-up. J Cachexia Sarcopenia Muscle. 2016 Sep;7(4):422-35. doi: 10.1002/jcsm.12091. Epub 2015 Dec 4. PMID 27239405
- [Result] Kho W, von Haefen C, Paeschke N, Nasser F, Endesfelder S, Sifringer M, Gonzalez-Lopez A, Lanzke N, Spies CD. Dexmedetomidine Restores Autophagic Flux, Modulates Associated microRNAs and the Cholinergic Anti-inflammatory Pathway upon LPS-Treatment in Rats. J Neuroimmune Pharmacol. 2022 Jun;17(1-2):261-276. doi: 10.1007/s11481-021-10003-w. Epub 2021 Aug 6. PMID 34357471
- [Result] Aranake-Chrisinger A, Avidan MS. Postoperative delirium portends descent to dementia. Br J Anaesth. 2017 Aug 1;119(2):285-288. doi: 10.1093/bja/aex126. No abstract available. PMID 28854545
- [Result] Peden CJ, Miller TR, Deiner SG, Eckenhoff RG, Fleisher LA; Members of the Perioperative Brain Health Expert Panel. Improving perioperative brain health: an expert consensus review of key actions for the perioperative care team. Br J Anaesth. 2021 Feb;126(2):423-432. doi: 10.1016/j.bja.2020.10.037. Epub 2021 Jan 4. PMID 33413977
- [Result] Jin Z, Hu J, Ma D. Postoperative delirium: perioperative assessment, risk reduction, and management. Br J Anaesth. 2020 Oct;125(4):492-504. doi: 10.1016/j.bja.2020.06.063. Epub 2020 Aug 11. PMID 32798069
- [Result] Meara JG, Leather AJ, Hagander L, Alkire BC, Alonso N, Ameh EA, Bickler SW, Conteh L, Dare AJ, Davies J, Merisier ED, El-Halabi S, Farmer PE, Gawande A, Gillies R, Greenberg SL, Grimes CE, Gruen RL, Ismail EA, Kamara TB, Lavy C, Lundeg G, Mkandawire NC, Raykar NP, Riesel JN, Rodas E, Rose J, Roy N, Shrime MG, Sullivan R, Verguet S, Watters D, Weiser TG, Wilson IH, Yamey G, Yip W. Global Surgery 2030: evidence and solutions for achieving health, welfare, and economic development. Int J Obstet Anesth. 2016 Feb;25:75-8. doi: 10.1016/j.ijoa.2015.09.006. Epub 2015 Sep 30. No abstract available. PMID 26597405
- [Result] Nijsse B, Visser-Meily JM, van Mierlo ML, Post MW, de Kort PL, van Heugten CM. Temporal Evolution of Poststroke Cognitive Impairment Using the Montreal Cognitive Assessment. Stroke. 2017 Jan;48(1):98-104. doi: 10.1161/STROKEAHA.116.014168. Epub 2016 Nov 29. PMID 27899753